CLINICAL TRIAL: NCT03237312
Title: The Impact of Serum Antimullerian Hormone Level on Adjusting the Number of Ovarian Drills in Polycystic Ovarian Syndrome
Brief Title: Serum Anti-mullerian Hormone and Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMH-PCOS
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Anti-Mullerian Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Other): Four punctures in each ovary were done regardless of the level of antimullerian hormone
  Interventions: Procedure: Laparoscopic ovarian drilling; Biological: Antimullerian hormone
- The study group (Other): The number of ovarian drills was adjusted according to antimullerian hormone level
  Interventions: Procedure: Laparoscopic ovarian drilling; Biological: Antimullerian hormone

INTERVENTIONS:
Procedure: Laparoscopic ovarian drilling — The electric current used was set at 40 Watts. The power was activated just before touching the ovary, and then the needle electrode was held against the antimesenteric surface of the ovary for 4 seconds until penetration of the ovarian capsule. Four or eight puncture points were made through the ovarian capsule of each ovary according to the study protocol. The ovaries were cooled in the pool of the Ringer's lactate after each cauterization both to minimize adhesion formation and to prevent heat trauma to the adjacent viscera. Complete hemostasis was ensured. At the end of the procedure, the ovaries were copiously rinsed with Ringer's lactate (Aqua-purator, Storz, Germany). An amount about 200 ml of heparinized Ringers lactate (5000 IU/1000 ml) was left in the pelvis to avoid postoperative adhesions.
Biological: Antimullerian hormone — 1. In patients with Antimullerian hormone between 4-8 ng/ml 4 punctures in each ovary were performed.
  2. In patients with Antimullerian hormone above 8 ng/ml 8 punctures in each ovary were performed.

SUMMARY:
In 1935 the polycystic ovary syndrome was a clinical diagnosis made on the morphological appearance of the ovaries in association with amenorrhoea, hirsutism and frequently obesity. At that time wedge resection of the ovaries was introduced on an empirical basis and proved a successful treatment for the associated anovulation and infertility. In the ensuing fifty years the limitations of a purely surgical approach to therapy have become recognized and the importance of the biochemical abnormalities appreciated. Prevalence of polycystic Ovary Syndrome: The prevalence of polycystic ovary syndrome in any specified population is dependent upon the diagnostic criteria used, but does have some regional and ethnic variation. While most reports on the prevalence of polycystic ovary syndrome range between 2 and 20%, the chosen diagnostic criteria are recognized to influence the determined prevalence. Anti-mullerian hormone which is a predictor of ovarian reserve is known to decrease after laparoscopic ovarian drilling. On the best of our knowledge no study had been done to use the level of anti-mullerian hormone as a factor for planning the number of ovarian drills in each ovary.

ELIGIBILITY:
Inclusion Criteria:

1. Infertility more than 2 years.
2. Age between 20-35 years.
3. clomiphene resistant patients: Patients received clomiphene 150 mg from day 3 to 7 of the menstrual cycle for 6 months and non-ovulatory (with failure of conception). They were followed up in the outpatient clinic.
4. No contraindications for laparoscopy.
5. Normal Hysterosalpingography

Exclusion Criteria:

1. Contraindications for laparoscopy e.g cardiac diseases, bad scared abdomen ect….
2. Women's age less than 20 years or more than 35 years.
3. Previous Laparoscopic surgery.
4. Previous ovarian surgery.
5. Women with Antimullerian hormone level less than 4 ng/ml.
6. Tubal factor infertility as diagnosed by Hysterosalpingography .

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Size of ovarian follicle (mm) | 14 days

SECONDARY OUTCOMES:
Antimullerian hormone level (ng/dl) | 3 months
Ovarian volume (ml) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided